CLINICAL TRIAL: NCT07094243
Title: Motivational Psychotherapy for Adolescent Depression and Academic Self-Concept: A Pilot Trial in a Non-Western Context
Brief Title: Motivational Psychotherapy for Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atefe Momeni (Other)
Responsible Party: Sponsor-Investigator, Atefe Momeni, Clinical Psychology Researcher, Islamic Azad University, Tehran Electronic Branch, Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Momeni2025-MP
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Depression; Low Academic Self-Concept
Keywords: Adolescent mental health; Motivational psychotherapy; Motivational interviewing; Academic self-concept; Pilot trial; Non-Western context
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Two parallel groups: a motivational psychotherapy group and a control group (no intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Psychotherapy (Experimental): Participants receive Motivational Psychotherapy intervention.
  Interventions: Behavioral: Motivational Psychotherapy
- No Intervention (No Intervention): Participants receive no psychological intervention during the study period.

INTERVENTIONS:
Behavioral: Motivational Psychotherapy — A structured short-term intervention based on motivational psychotherapy, delivered in individual sessions over 8 weeks to improve adolescent depression and academic self-concept.
  Arms: Motivational Psychotherapy

SUMMARY:
This pilot study investigates the effectiveness of Motivational Psychotherapy in reducing symptoms of depression and improving academic self-concept among adolescent girls in Iran. A total of 30 participants aged 13 to 17 were randomly assigned to an experimental group receiving Motivational Psychotherapy and a control group receiving no treatment. The intervention consisted of 8 weekly sessions based on the principles of motivational interviewing and was tailored to adolescent needs. Outcomes were measured using the Beck Depression Inventory-II (BDI-II) and the Academic Self-Concept Questionnaire (ASCQ). Results suggest the potential benefit of this culturally sensitive approach in non-Western adolescent populations.

DETAILED DESCRIPTION:
This randomized controlled pilot trial evaluated the effectiveness of Motivational Psychotherapy in reducing depressive symptoms and improving academic self-concept among adolescent girls in Iran. A total of 30 participants aged 13-17 years were randomly assigned to either the Motivational Psychotherapy group or a no-intervention control group.

The intervention consisted of 8 weekly individual sessions (60 minutes each) based on a manualized Motivational Psychotherapy protocol, adapted for adolescents in a non-Western context. The sessions focused on resolving ambivalence, enhancing intrinsic motivation, and strengthening environmental support.

Outcome measures included the Beck Depression Inventory-II (BDI-II) for depressive symptoms and the Academic Self-Concept Questionnaire (ASCQ) for academic self-concept. Data were analyzed using ANCOVA to control for baseline differences between groups. The results showed significant improvement in depression scores and academic self-concept in the intervention group compared to the control group, supporting the feasibility and cultural relevance of Motivational Psychotherapy for adolescent mental health.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Female adolescents aged 13 to 17 years
* Clinical diagnosis of mild to moderate depression based on DSM-5 criteria
* Currently enrolled in middle or high school
* Informed consent obtained from parents/legal guardians and assent from adolescents

Exclusion Criteria:

* Severe depression requiring urgent psychiatric care
* Diagnosis of a major psychiatric disorder (e.g., bipolar disorder, psychosis)
* Ongoing psychotherapy or psychotropic medication use
* Significant cognitive or developmental disability interfering with participation

Exclusion Criteria:

-

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Depression Score from Baseline to 8 Weeks Post-Intervention | Baseline and 8 weeks after start of intervention
  Depression symptoms will be assessed using the Beck Depression Inventory-II (BDI-II; range 0-63, higher scores indicate worse depression). The mean change in BDI-II scores from baseline to 8 weeks will be analyzed between the Motivational Psychotherapy and control groups.

SECONDARY OUTCOMES:
Change in Depression Score from Baseline to 8 Weeks Post-Intervention | Baseline and 8 weeks after start of intervention
  Depression symptoms will be assessed using the Beck Depression Inventory-II (BDI-II). The primary outcome is the mean change in BDI-II scores from baseline to 8 weeks after the intervention. The comparison will be made between the experimental group (receiving motivational psychotherapy) and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Sahebdel, Associate Professor of Counsel, Principal Investigator — Islamic Azad University, Tehran Electronic Branch
Locations (1):
- Islamic Azad University, Tehran Electronic Branch, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effectiveness of Motivational Psychotherapy in Adolescent Depression — https://doi.org/10.18502/htaa.v7i3.14214